CLINICAL TRIAL: NCT01000623
Title: Evaluation of a Biobehavioral Intervention for Hot Flashes
Brief Title: Venlafaxine and Hypnosis or Focused Attention in Treating Patients with Hot Flashes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MC09C7; NCI-2009-01303 (Registry Identifier: NCI's CTRO); 09-003233 (Other: Mayo Clinic IRB); MC09C7 (Other: Mayo Clinic Cancer Center)
Record Dates: First submitted 2009-10-19; First posted 2009-10-23 (Estimated); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Hot Flashes
MeSH Terms: conditions — Hot Flashes | interventions — Venlafaxine Hydrochloride; Hypnosis; Mind-Body Therapies

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm I (Experimental): Patients receive oral venlafaxine once or twice daily in weeks 2-8. Patients see a therapist once a week to learn hypnosis in weeks 2-5. Patients continue hypnosis at home in weeks 6-8.
  Interventions: Drug: venlafaxine; Procedure: hypnotherapy
- Arm II (Active Comparator): Patients receive oral venlafaxine once or twice daily in weeks 2-8. Patients see a therapist once a week to learn focused attention in weeks 2-5. Patients continue focused attention at home in weeks 6-8.
  Interventions: Drug: venlafaxine; Procedure: mind-body intervention procedure
- Arm III (Active Comparator): Patients receive oral placebo once or twice daily in weeks 2-8. Patient see a therapist once a week to learn hypnosis in weeks 2-5. Patients continue hypnosis at home in weeks 6-8.
  Interventions: Drug: placebo; Procedure: hypnotherapy
- Arm IV (Active Comparator): Patients receive oral placebo once or twice daily in weeks 2-8. Patient see a therapist once a week to learn focused attention in weeks 2-5. Patients continue focused attention at home in weeks 6-8.
  Interventions: Drug: placebo; Procedure: mind-body intervention procedure

INTERVENTIONS:
Drug: venlafaxine — Given orally
  Other Names: Effexor; VNF
  Arms: Arm I; Arm II
Drug: placebo — Given orally
  Other Names: PLCB
  Arms: Arm III; Arm IV
Procedure: hypnotherapy — Practice hypnosis
  Other Names: hypnosis
  Arms: Arm I; Arm III
Procedure: mind-body intervention procedure — Practice focused attention
  Other Names: mind-body interventions
  Arms: Arm II; Arm IV

SUMMARY:
Rationale: Venlafaxine may help relieve hot flashes in women who have had breast cancer. Hypnosis or focused attention may help control hot flashes in postmenopausal women. It is not yet known whether giving venlafaxine together with hypnosis or focused attention is more effective in treating hot flashes.

Purpose: This randomized clinical trial is studying venlafaxine together with hypnosis or focused attention in treating patients with hot flashes.

DETAILED DESCRIPTION:
Objectives:

I. To evaluate the effect of hypnosis plus venlafaxine versus focused attention with venlafaxine versus hypnosis plus a placebo versus focused attention plus a placebo for reducing hot flashes.

II. To evaluate the side effects associated with hypnosis with venlafaxine versus focused attention with venlafaxine versus hypnosis plus a placebo versus focused attention plus a placebo for reducing hot flashes.

III. To evaluate the effects of the four treatment arms on mood, sleep, hot flash interference and menopause quality of life.

IV. To explore the role of expectancy and hypnotizability as moderators of the effect of each of the four treatment arms in reducing hot flashes.

Outline: Patients are randomized to 1 of 4 intervention arms. Patients receive oral venlafaxine or a placebo and practice hypnosis or focused attention.

ELIGIBILITY:
Inclusion

* Women with a history of breast cancer (currently without malignant disease) or women who have no history of breast cancer but who wish to avoid estrogen due to a perceived increased risk of breast cancer
* Women over the age of 18 who are postmenopausal and wish to avoid hormonal therapy to treat menopausal symptoms
* Postmenopausal as defined by:

  1. no menstrual period in the past 12 months;
  2. no menstrual period in the past 6 months and an FSH level greater than 40; or
  3. women who have had a bilateral oophorectomy
* If women have had a hysterectomy and still have their ovaries, they must meet the FSH criteria described above
* Note: We are excluding women of childbearing potential as this is a pilot trial and allowing women of childbearing potential with hot flashes to participate would introduce a hormonal heterogeneous population that would confound the ability to answer the research question
* Bothersome hot flashes (defined by their occurrence >= 28 times per week [about 4 per day]) and of sufficient severity to make the patient desire therapeutic intervention
* Presence of hot flashes for >=1 month prior to study entry
* Life expectancy >= 6 months
* ECOG Performance Status (PS) 0 or 1
* Possession of a CD/DVD player or ability to play a CD Exclusion
* Any of the following current (=< last 4 weeks) or planned therapies: antineoplastic chemotherapy, androgens, estrogens, progestational agents, other herbal supplements, including soy (herbal teas from a store are allowed), or Warfarin (1 mg of daily warfarin is allowed for central line patency)
* Tamoxifen, raloxifene, or aromatase inhibitors are allowed, but the patient must have been on a constant dose for >= 4 weeks and ust not be expected to stop the medication during the study period
* History of allergic or other adverse reaction to venlafaxine or SSRI's
* Current or planned use of other agents for treating hot flashes
* Use of venlafaxine or hypnosis in the past 6 months
* Diagnosis of/problems with chronic diarrhea or history of bowel obstruction or esophageal stricture
* Pregnant women or nursing women
* Current or planned use of any type of antidepressants
* Diagnosis of major depressive episode, acute anxiety disorder, liver or kidney dysfunction (defined by SGOT and creatinine levels 1.5 x upper limit of normal) as listed in the patient's medical history in the chart within the past year and by self report
* Uncontrolled hypertension (defined as 3 consecutive readings over the past year of over 160 systolic, and over 100 diastolic)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2010-01-31 (Actual); Primary Completion 2012-02-28 (Actual); Study Completion 2015-09-08 (Actual)

PRIMARY OUTCOMES:
Hot flash score measured by hot flash diary data | Baseline
Hot flash severity measured by hot flash diary data | Baseline
Hot flash frequency measured by hot flash diary data | Baseline
Hot flash score measured by hot flash diary data | Daily during study, weeks 2-8
Hot flash severity measured by hot flash diary data | Daily during study, weeks 2-8
Hot flash frequency measured by hot flash diary data | Daily during study, weeks 2-8

SECONDARY OUTCOMES:
Side effects measured by CTCAE v 3.0 and patient reports | Baseline
Side effects measured by CTCAE v 3.0 and patient reports | Once a week, weeks 2-8
Sleep effects measured by Modified Medical Outcomes Sleep Scale questionnaire | Baseline
Mood measured by Profile of Mood States questionnaire | Baseline
Menopause quality of life measured by MENQOL questionnaire | Baseline
Daily interference measured by Hot Flash Related Daily Interference Scale questionnaire | Baseline
Sleep effects measured by Modified Medical Outcomes Sleep Scale questionnaire | Week 8
Mood measured by Profile of Mood States questionnaire | Week 8
Menopause quality of life measured by MENQOL questionnaire | Week 8
Daily interference measured by Hot Flash Related Daily Interference Scale questionnaire | Week 8
Evaluate the moderating effect of the expectations for the intervention to be effective and the ability of the person to be hypnotized | Week 5

CONTACTS AND LOCATIONS:
Overall Officials: Debra L. Barton, R.N., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States